CLINICAL TRIAL: NCT06389838
Title: Prospektiv Randomisierte Studie Zur Multimodalen Selbstbehandlung Von Frauen Mit Inkontinenzbeschwerden Mit Einer Digitalen Gesundheitsanwendung
Brief Title: RCT on Multimodal Self-treatment for Women With Incontinence Using a Digital Health Application
Acronym: DINKS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kranus Health GmbH (Industry)
Collaborators: Johannes Gutenberg University Mainz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DINKS01; DRKS00033704 (Registry Identifier: DRKS); 2024-512094-27 (EudraCT Number)
Record Dates: First submitted 2024-04-25; First posted 2024-04-29 (Actual); Results first posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Urinary Incontinence,Stress; Urinary Incontinence, Urge; Urinary Incontinence; Overactive Bladder Syndrome; Female Urinary Stress Incontinence
Keywords: Urinary Incontinence; Mobile Health; Digital therapeutics; Pelvic Floor exercises; bladder control; digital health; app based therapy; behavioral intervention; quality of life
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence, Urge; Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, controlled, single-blinded, 2-arm design
Who Masked: Investigator
Masking Description: Participants know which group they are assigned to, but the investigators are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention through a digital therapy program aimed at multimodal self-treatment for incontinence in addition to standard of care
  Interventions: Device: Kranus Mictera
- Control (No Intervention): Participants will continue with their therapy treatment (standard of care) if they are on it for more that four weeks before inclusion. Beginning of new therapies during the study is not allowed.

INTERVENTIONS:
Device: Kranus Mictera — An app-based digital therapy program aimed at multimodal self-treatment for incontinence. The app is certified class I medical device (MDR).
  Arms: Intervention

SUMMARY:
This study, titled "Prospective Randomized Study on Multimodal Self-Treatment for Women with Incontinence Symptoms Using a Digital Health Application," abbreviated as DINKS, aims to investigate the efficacy of a digital health application in treating incontinence in women. The study involves a single-center, single blinded, randomized, controlled trial with two arms: one receiving digital therapy intervention and the other serving as a control group with standard of care. The primary objective is to reduce the frequency of incontinence episodes over a 12-week intervention period, with secondary goals including improvements in disease symptoms, quality of life, and patient activation. The study plans to recruit 198 female participants and assess various endpoints related to incontinence severity, quality of life, and treatment outcomes.

DETAILED DESCRIPTION:
The intervention in this study involves a digital therapy program delivered via a smartphone or tablet application. This program includes several components aimed at addressing different aspects of incontinence management:

Voiding Diary: Participants will be instructed to maintain a diary to track their urinary habits, including frequency of voiding, episodes of incontinence, and fluid intake.

Pelvic Floor Exercises and Physiotherapy: The digital therapy program will provide guidance on performing pelvic floor exercises and other physiotherapeutic interventions aimed at strengthening pelvic floor muscles and improving bladder control.

Bladder Training and Cognitive Behavioral Therapy: Participants will receive instructions on bladder training techniques and cognitive behavioral strategies to manage urgency and frequency of urination.

Mental Exercises: The program will include mental exercises such as mindfulness techniques, progressive muscle relaxation, and stimulus control methods to help participants manage stress, anxiety, and other psychological factors contributing to incontinence.

Acute Urgency Management: Strategies for managing acute episodes of urgency and urge incontinence will be provided, including techniques to delay voiding and control bladder spasms.

Educational and Nutritional Guidance: Participants will have access to educational materials and nutritional guidance aimed at optimizing bladder health and overall well-being.

Progress Tracking and Motivation: The application will feature tools for tracking progress, setting goals, and providing motivational feedback to encourage adherence to the intervention.

Overall, the digital therapy program is designed to provide comprehensive support for women with incontinence symptoms, addressing both physical and psychological aspects of the condition to improve symptom severity, quality of life, and patient activation.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years or older.
* Diagnosis of urinary incontinence, including stress incontinence, urge incontinence, or mixed incontinence.
* Mastery of the German language.
* Access to the internet.
* Access to a tablet or smartphone (Android not older than version 7 and iPhone not older than iPhone 9).
* Ability to provide informed consent

Exclusion Criteria:

* Acute cystitis (N30.0)
* Bladder stones (N21.0)
* Recurrent, uncontrollable macrohematuria (R31)
* Newly diagnosed bladder carcinoma < 3 months (C67)
* Relative Exclusion Criteria not coded according to ICD-10:
* Inability to physically participate in the therapy program
* Active pregnancy
* Bladder botulinum toxin treatment within the last 6 months
* Study-specific methodological exclusion criteria:
* Patients unable to understand and independently sign the consent form
* Initiation of new medication or physical therapy for urinary symptoms within the last 4 weeks
* Severe psychiatric disorders hindering app usage
* Neurological disorders affecting the urinary tract
* Incontinence or tumor surgeries in the pelvic area
* Severe obesity (BMI >35)
* Recurrent urinary tract infections (at least 2 within 6 months or 3 within a year)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2024-04-30 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Axel Haferkamp, PhD, Principal Investigator — Director of the Clinic of Urology, University of Mainz , Germyny
Locations (1):
- Clinic of Urology, Mainz, Germany

IPD SHARING:
Plan to Share IPD: No
Study protocol and study report will be shared

REFERENCES:
- [Derived] Haferkamp A, Frey L, Duwe G, Borner JH, Hunfeld C, Brocker KA, Troilo S, Lehmacher W, Papp CP, Miller K, Wiemer L. App-based therapy for female patients with urinary incontinence in Germany (DINKS): a single-blind, randomised, controlled trial. Lancet Digit Health. 2025 Dec;7(12):100935. doi: 10.1016/j.landig.2025.100935. Epub 2025 Dec 16. PMID 41407582
- See also: Kranus webpage for the medical device — https://kranushealth.com/de/fachkreise/mictera

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Participants will continue their therapy treatment (standard of care) if they are on it for more than four weeks before inclusion.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 96 | 98
Completed | 92 | 94
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 96 | 98 | 194
Age, Continuous [Median (Standard Deviation); unit: years] | 48.5 (11.65) | 51.0 (12.01) | 50.0 (11.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 98 | 194
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 96 | 98 | 194
BMI [Mean (Standard Deviation); unit: kg/m2] | 25.04 (4.11) | 25.69 (4.47) | 25.37 (4.24)
Type of incontinence [Count of Participants; unit: Participants] — Population: Proportion of participants with either stress, urge and mixed incontinence.
  Participants
    Stress incontinence | 60 | 61 | 121
    Urge incontinence | 21 | 22 | 43
    Mixed incontinence | 15 | 15 | 30
Duration of incontinence [Mean (Standard Deviation); unit: year] | 5.31 (6) | 5.21 (5.55) | 5.26 (5.76)
Number of incontinence episodes per 24h [Mean (Standard Deviation); unit: episodes] | 3.71 (2.32) | 3.57 (2.09) | 3.64 (2.2)
Country of birth [Count of Participants; unit: Participants]
  Germany | 82 | 88 | 170
  Russian Federation | 3 | 3 | 6
  United Kingdom | 1 | 1 | 2
  Kyrgyzstan | 2 | 0 | 2
  Others | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Incontinence Episodes
Description: Relative change (rel-CfB-IEF) of IEF from baseline to week 12 relative to baseline; desired reduction in mean relative IEF by 50%; IEF per 24 hours - averaged over 72 hours.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: number of incontinencies
Arm/Group | Intervention | Control
Number analyzed (Participants) | 96 | 98
number of incontinencies | -2.25 (2.26) | -0.14 (1.45)

2. Secondary Outcome: International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF)
Description: ICIQ-SF assess the frequency and severity of urinary incontinence and its impact on the quality of life of those affected.
  Score range: 0 - 21 points, with higher values representing a worse outcome. Outcome measure: change in ICIQ-SF from baseline to week 12.
Time Frame: 12 weeks
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 96 | 98
scores on a scale | -3.94 [-12 to 3] | -0.27 [-7 to 4]

3. Secondary Outcome: Incontinence Quality-of-Life (I-QOL)
Description: I-QoL assesses the impact of urinary incontinence on quality of life. Scale score ranging from 0-100. Higher scores on the I-QOL indicate a better quality of life, while lower scores indicate greater impairment due to urinary incontinence.
  Outcome measure: change in I-QoL from baseline to week 12.
Time Frame: 12 weeks
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 96 | 98
scores on a scale | 17.9 [-24 to 65] | 1.16 [-30 to 27]

4. Secondary Outcome: Patient Activation Measure-13 (PAM-13)
Description: The PAM-13 assesses patients' self-competence and knowledge about their own health.
  The range is from 0 to 100 points, with higher scores for a higher level of activation.
  Outcome Measure: Change in PAM-13 score from baseline to week 12.
Time Frame: 12 weeks
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 96 | 98
scores on a scale | 7.35 [-73 to 58] | 0.51 [-14 to 43]

5. Secondary Outcome: Patient Global Impression of Improvement (PGI-I)
Description: The PGI-I is a subjective assessment of the improvement in state of health or symptoms. It consists of a single question that asks patients to give their own assessment of the improvement in their state of health.
  Scale: from "much better" to "much worse". Outcome measure: Count of participants who had an improvement ("minimally better" or higher) in PGI-I value at week 12.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 92 | 94
Participants | 84 | 11

6. Secondary Outcome: Cured Patients
Description: Proportion of patients without incontinence (cured patients) at study end
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 96 | 98
Participants | 22 | 2

7. Secondary Outcome: Urinary Frequency Day
Description: Change in urinary frequency during the day from baseline to week 12. The outcome measure was assessed via the optional app diary, so data was available only for intervention group users who utilized this feature.
Time Frame: 12 weeks
Population: Data was available only for intervention group users who utilized this feature, leaving the control group without corresponding data. Entry was optional for the participants using the app. Therefore, there is a lower number of participant for this analysis.
Measure: Mean (Standard Deviation); unit: urination events per day
Arm/Group | Intervention
Number analyzed (Participants) | 66
urination events per day | -1.51 (2.28)

8. Secondary Outcome: Urinary Frequency Night
Description: Change in urinary frequency at night from baseline to week 12. The outcome measure was assessed via the optional app diary, so data was available only for intervention group users who utilized this feature.
Time Frame: 12 weeks
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: urination events per night
Groups:
- Intervention Group: Intervention through a digital therapy program aimed at multimodal self-treatment for incontinence in addition to standard of care
Arm/Group | Intervention Group
Number analyzed (Participants) | 39
urination events per night | -0.29 (0.62)

9. Secondary Outcome: Pad Use
Description: Change in pad use from baseline to week 12
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: pads
Arm/Group | Intervention | Control
Number analyzed (Participants) | 96 | 98
pads | -2.63 (4.37) | 0.15 (3.50)

10. Secondary Outcome: Urge Incontinence
Description: Change in urge incontinence from baseline to week 12. The outcome measure was assessed via the optional app diary, so data was available only for intervention group users who utilized this feature.
Time Frame: 12 weeks
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: episodes
Arm/Group | Intervention
Number analyzed (Participants) | 14
episodes | -0.84 (1.82)

11. Secondary Outcome: Functional Bladder Capacity
Description: Change in functional bladder capacity from baseline to week 12. The outcome measure was assessed via the optional app diary, so data was available only for intervention group users who utilized this feature.
Time Frame: 12 weeks
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Intervention
Number analyzed (Participants) | 66
ml | 48.28 (57.48)

12. Secondary Outcome: Number of Participants With Treatment Failure
Description: Proportion of patients with treatment failure within the study period, defined as any reported worsening in the PGI-I questionnaire at the end of the study or the start of any interventions against the incontinence symptoms (conservative and invasive methods).
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 96 | 98
Participants | 4 | 20

13. Secondary Outcome: Stress Urinary Incontinence Episodes of the S/U-IQ
Description: Change in stress urinary incontinence episodes of the S/U-IQ
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: episodes
Arm/Group | Intervention | Control
Number analyzed (Participants) | 96 | 98
episodes | -10.14 (14.69) | -0.59 (12.94)

14. Secondary Outcome: Urgency Urinary Incontinence Episodes of the S/U-IQ
Description: Change in urgency urinary incontinence episodes of the S/U-IQ
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: eisodes
Arm/Group | Intervention | Control
Number analyzed (Participants) | 96 | 98
eisodes | -1.53 (11.13) | 0.67 (7.89)

ADVERSE EVENTS:
Time Frame: For an average of 3 months.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/96 | 0/98
Serious Adverse Events (participants affected / at risk) | 0/96 | 0/98
Other Adverse Events (participants affected / at risk) | 0/96 | 0/98

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-14): https://cdn.clinicaltrials.gov/large-docs/38/NCT06389838/Prot_SAP_000.pdf